CLINICAL TRIAL: NCT00843531
Title: A Phase II Study to Evaluate the Safety and Efficacy of RAD001 Plus Erlotinib in Patients With Well- to Moderately-Differentiated Neuroendocrine Tumors
Brief Title: RAD001 and Erlotinib in Patients With Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry); Novartis Pharmaceuticals (Industry); The V Foundation for Cancer Research (Other)
Responsible Party: Principal Investigator, Emily Bergsland, Sponsor-Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 084511; NCI-2011-01291 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine; islet cell; carcinoid; pancreatic neuroendocrine; paraganglioma; pheochromocytoma; RAD001; everolimus; erlotinib; Tarceva
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Paraganglioma; Pheochromocytoma | interventions — Everolimus; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAD001 and erlotinib (Experimental): Each 28 day cycle:
  RAD001: 5 mg per day by mouth (self-administered) Erlotinib: 100 mg per day by mouth (self-administered)
  Interventions: Drug: RAD001; Drug: erlotinib

INTERVENTIONS:
Drug: RAD001 — 5 mg/day PO (oral)
  Other Names: Everolimus
Drug: erlotinib — 100 mg/day (oral)
  Other Names: Tarceva

SUMMARY:
The purpose of this study is to test how safe and effective the combination of RAD001 and erlotinib is in patients with neuroendocrine tumors.

DETAILED DESCRIPTION:
Preclinical data suggest that concomitant inhibition of two non-redundant amplified pathways (mTOR and EGFR) can reverse drug resistance and more profoundly affect tumor growth than targeting either pathway alone. EGFR inhibitors may abrogate feedback loops that stimulate upstream signaling events such as PI3K and Akt in the face of mTOR inhibition. Although ErbB receptors signal through mTOR-dependent mechanisms, mTOR-independent ErbB receptor signaling also occurs in cancer. Furthermore, deregulation of apoptotic pathways like the PI3K/Akt/PTEN axis (e.g. via PTEN loss of function or AKT gene amplification) may lead to resistance to EGFR inhibitors. Treatment with an inhibitor of mTOR may reverse this resistance. Targeting the mTOR and EGFR pathways concurrently may more effectively inhibit tumor growth than inhibiting either pathway alone.

The compelling preclinical data, coupled with modest single agent activity seen with EGFR inhibition and mTOR inhibition in neuroendocrine tumors (NETs), provides a strong rationale for studying the activity of concomitant pathway inhibition in patients with advanced NETs. Support for this strategy also stems from the fact that EGFR inhibitors can be safety combined with mTOR inhibitors in humans. Emerging data from a phase I study of RAD001 plus erlotinib in patients with previously treated advanced non-small cell lung cancer (NSCLC) suggests that the two agents can be safely combined at the following doses: RAD001 5 mg PO q D and erlotinib 150 mg PO qD.

Of note, the original dose selections for RAD001 and erlotinib for this study stem directly from phase I studies with this combination (RAD001 5 mg PO qD plus erlotinib 150 mg PO qD). The modified dose selections (RAD001 5 mg PO qD plus erlotinib 100 mg PO qD) are the result of integrating discussions with the study sponsor, preliminary safety data from the first few patients enrolled in this study (suggesting that some patients tolerate full-dose therapy and others do not) and additional phase I data suggesting that the maximum tolerated dose (MTD) in some patient populations is lower than in others, e.g. the MTD in breast cancer patients is RAD001 2.5 mg PO qD and erlotinib 100 mg PO QD (Mayer et al. American Society of Clinical Oncology (ASCO) 2009 Breast Cancer Symposium, Abstract #254).

ELIGIBILITY:
Inclusion Criteria:

* >=1 measurable disease site per RECIST, not previously irradiated (if previous radiation to marker lesion(s), need evidence of PD)
* Histologic dx of well- to moderately-differentiated NET: low- or intermediate-grade, islet cell carcinoma, pancreatic NET, carcinoid, atypical carcinoid, paraganglioma, pheochromocytoma. No longer enrolling carcinoid patients as of 4/25/2011.
* ≥4 wks since completion of prior investigational drug tx or other tx(radiation, chemotherapy, immunotherapy, antibody-based tx); recovery from acute toxicities of prior tx
* Eastern Cooperative Oncology Group (ECOG) ≤2
* Absolute Neutrophil Count (ANC) ≥1500/μL
* Plts ≥100,000/μL
* Hgb >9 gm/dL
* Total bilirubin ≤2.0 mg/dL or 1.5X upper limit of normal (ULN)
* Serum transaminases ≤2.5x ULN (≤5xULN if liver mets)
* Serum Cr ≤2.0 mg/dL or 1.5X ULN
* Fasting serum glucose <150 mg/dL or <1.5x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤2.5xULN
* International Normalized Ratio (INR) ≤1.5
* Written informed consent, compliance w/study requirements
* Archived tissue if available
* Negative urine/serum pregnancy test w/in 7 days prior to Day 1

Exclusion Criteria:

* Poorly differentiated NET, high-grade NET, adenocarcinoid, goblet cell carcinoid, small cell carcinoma
* Major surgery or traumatic injury w/in 4 wks, inadequate recovery from side effects of any surgery, or likely to require major surgery during study
* Liver-directed therapy w/in 2 mths of enrollment. Prior tx w/ radiotherapy (including radiolabeled spheres, cyberknife, hepatic arterial embolization (w/ or w/o chemotherapy), cryotherapy/ablation) allowed if areas of measurable disease being used for the study are not affected, or if PD can clearly be documented in the area
* Prior tx w/ EGFR inhibitor or mTOR inhibitor
* Known hypersensitivity to RAD001 or other rapamycins
* Chronic, systemic tx w/ corticosteroids or another immunosuppressive agent (topical or inhaled corticosteroids are allowed)
* Immunization w/ attenuated live vaccines w/in 1 wk of study entry or during study
* Uncontrolled brain or leptomeningeal mets, including pts who continue to require glucocorticoids for brain or leptomeningeal mets
* Other malignancies w/in the past 3 years except for adequately treated carcinoma of the cervix, basal/squamous cell skin carcinomas, or other in situ cancer
* Severe and/or uncontrolled intercurrent medical conditions or other conditions that may affect study participation, including, but not limited to:
* Severely impaired lung function (spirometry and Diffusing capacity of the lungs for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or O2 saturation ≤88% at rest on room air)
* Symptomatic congestive heart failure (CHF) of New York Heart Association (NYHA) Class III or IV
* Unstable angina pectoris, symptomatic CHF, myocardial infarction w/in 6 months of Day 1, uncontrolled cardiac arrhythmia or any other significant cardiac disease
* Uncontrolled diabetes (fasting serum glucose ≥ 150 mg/dL or >1.5x upper limit of normal (ULN))
* Any active (acute or chronic) or severe infection, disorder, or nonmalignant medical illness that is uncontrolled or whose control may be jeopardized by study tx
* Liver disease
* Hx of HIV seropositivity or other immunocompromised state
* GI function impairment or disease that may alter absorption of RAD001 or erlotinib
* Active, bleeding diathesis or on oral anti-vitamin K medication (patients needing anticoagulation must use low molecular weight heparin (LMWH))
* Hx of other disease, metabolic dysfunction, or physical exam or lab finding giving reasonable suspicion of disease/condition that contraindicates study tx, might affect study results or puts the pt at high risk
* Pregnant or breast feeding females
* Adults of reproductive potential not willing to use effective methods of birth control during tx and ≥8 wks after completing tx
* Inability to comply w/ objectives and procedures
* Inability to comply w/ concomitant medication restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-06-25 (Actual); Primary Completion 2013-07-16 (Actual); Study Completion 2016-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Bergsland, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001 and Erlotinib: RAD001 and erlotinib
  Each 28 day cycle:
  RAD001: 5 mg per day by mouth (self-administered) Erlotinib: 100 mg per day by mouth (self-administered)
Period: Overall Study
Arm/Group | RAD001 and Erlotinib
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- RAD001 and Erlotinib: * everolimus 5 mg daily and continued this throughout the duration of treatment
  * erlotinib at a dose of 100 mg daily with the option to dose reduce erlotinib to 100 mg daily in the setting of grade 3/4 rash or diarrhea
  * cycles defined as every 28 days
Arm/Group | RAD001 and Erlotinib
Number analyzed (Participants) | 17
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1
  30-39 years | 0
  40-49 years | 2
  50-59 years | 2
  60-69 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Neuroendocrine Tumor Type [Count of Participants; unit: Participants]
  Carcinoid Neuroendocrine Tumor | 9
  Pancreatic neuroendocrine tumor (PNET) | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response is defined as complete response (CR) or partial response (PR) assessed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. The primary analysis population is based on efficacy-evaluable patients, defined as those patients who receive at least one cycle of RAD001 plus erlotinib and undergo at least one post-baseline response assessment or die while on therapy.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- RAD001 Plus Erlotinib: * everolimus 5 mg daily and continued this throughout the duration of treatment
  * erlotinib at a dose of 100 mg daily with the option to dose reduce erlotinib to 100 mg daily in the setting of grade 3/4 rash or diarrhea
  * cycles defined as every 28 days
Arm/Group | RAD001 Plus Erlotinib
Number analyzed (Participants) | 17
Participants | 0

2. Secondary Outcome: Number of Patients With Dose-limiting Toxicity (DLT)
Description: Primary safety analysis will be conducted after the first 16 patients have had potential for completion of two cycles of protocol therapy. All patients receiving at least one dose of protocol therapy will be included in the analyses. All patients with treatment-related, Grade 3 or higher adverse events according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3 resulting in a DLT will be reported.
Time Frame: Up to 9 months
Measure: Count of Participants; unit: Participants
Groups:
- RAD001 and Erlotinib: Each 28 day cycle:
  RAD001: 5 mg per day by mouth (self-administered) Erlotinib: 100 mg per day by mouth (self-administered)
  RAD001: 5 mg/day PO (oral)
  erlotinib: 100 mg/day (oral)
Arm/Group | RAD001 and Erlotinib
Number analyzed (Participants) | 17
Participants | 8

3. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response will be defined as the time from the initial documentation of response to documented disease progression or death from any cause on study
Time Frame: Up to 2 years
Measure: Number; unit: months
Arm/Group | RAD001 and Erlotinib
Number analyzed (Participants) | 17
months | NA — No participants obtained an objective response

4. Secondary Outcome: Overall Survival
Description: Overall survival will be defined as the time from first day of treatment until death
Time Frame: Up to 3 years
Population: Data for overall survival not collected
Arm/Group | RAD001 and Erlotinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: PFS will be defined as the time from the first day of treatment and documented objective response to time of progression or death from any cause, whichever occurs first
Time Frame: Up to 3 years
Population: No participants obtained an objective response (CR or PR) therefore data for long term progression-free survival data was not collected.
Arm/Group | RAD001 and Erlotinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Progression
Description: Time to disease progression will be defined as the time from baseline until documented disease progression or death (whichever occurs first).
Time Frame: Up to 3 years
Population: Data for time to progression not collected
Groups:
- RAD001 Plus Erlotinib: RAD001 and erlotinib
  Each 28 day cycle:
  RAD001: 5 mg per day by mouth (self-administered) Erlotinib: 100 mg per day by mouth (self-administered)
Arm/Group | RAD001 Plus Erlotinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time to treatment failure will be defined as the time from first day of treatment until study discontinuation (for any cause).
Time Frame: Up to 3 years
Population: Data for time to treatment failure not collected
Groups:
- Carcinoid Tumors: * everolimus 5 mg daily and continued this throughout the duration of treatment
  * erlotinib at a dose of 100 mg daily with the option to dose reduce erlotinib to 100 mg daily in the setting of grade 3/4 rash or diarrhea
  * cycles defined as every 28 days
Arm/Group | Carcinoid Tumors
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | RAD001 Plus Erlotinib
All-Cause Mortality (participants affected / at risk) | 6/17
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 Plus Erlotinib (N=17)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema: limb (Vascular disorders) | 1 (2)
Creatinine (Investigations) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Pain - Other - Right upper quadrant pain (Investigations) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 Plus Erlotinib (N=17)
Stomatitis (Gastrointestinal disorders) | 13 (41)
Diarrhea (Gastrointestinal disorders) | 15 (36)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 11 (24)
Anorexia (Metabolism and nutrition disorders) | 11 (14)
Fatigue (General disorders) | 13 (21)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (8)
Dry Skin (Skin and subcutaneous tissue disorders) | 11 (13)
Weight Loss (Investigations) | 9 (16)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Dysgeusia (Nervous system disorders) | 9 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (20)
Creatinine (Renal and urinary disorders) | 6 (15)
Nail changes (Skin and subcutaneous tissue disorders) | 6 (11)
Dehydration (Metabolism and nutrition disorders) | 6 (10)
Hypercholesteremia (Investigations) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 6 (8)
Hyponatremia (Metabolism and nutrition disorders) | 5 (11)
Flatulence (Gastrointestinal disorders) | 5 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 4 (11)
Edema: limb (Vascular disorders) | 4 (11)
Vomiting (Gastrointestinal disorders) | 4 (10)
Nausea (Gastrointestinal disorders) | 4 (9)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4 (7)
Pain - Head/headache (Nervous system disorders) | 4 (4)
Alkaline phosphatase (Investigations) | 3 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 (4)
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Cardiac disorders) | 3 (3)
Hemoglobin (Investigations) | 3 (3)
Chills (General disorders) | 3 (3)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 2 (12)
Lymphopenia (Blood and lymphatic system disorders) | 2 (4)
Cough (Reproductive system and breast disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2)
Platelets (Blood and lymphatic system disorders) | 2 (4)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (3)

LIMITATIONS AND CAVEATS:
Study was terminated earlier than expected due to insufficient efficacy at interim analysis and overall low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes